CLINICAL TRIAL: NCT06159088
Title: Improved Gut Health Outcomes Associated With Feihe Probiotics Fortified With Hydrolyzed Whey Protein in Infant Formula: A Randomized, Controlled Trial
Brief Title: Improved Gut Health Outcomes Associated With Probiotics Fortified With Hydrolyzed Whey Protein in Infant Formula
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heilongjiang Feihe Dairy Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 22-SM-11-FEIHE-003
Record Dates: First submitted 2023-11-26; First posted 2023-12-06 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Gut Health; Gastrointestinal Diseases
Keywords: Infant Formula; Prebiotics; Hydrolyzed Whey Protein
MeSH Terms: conditions — Gastrointestinal Diseases | interventions — Lactation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Two arms of participants will be assigned masked products (investigational formula and control formula) after randomization, while the participants of breastfeeding arm will not be assigned study products.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Feihe Investigational Formula (Experimental): Feihe Investigational Formula
  1. With the highest probiotic content
  2. Containing 2' -fucosyl lactose
  3. Add hydrolyzed whey protein
  4. Comprehensive nutrition: OPO, lactoferrin, CPP, nucleotide, choline, inositol, taurine, L-carnitine, GOS, lutein
  Interventions: Dietary Supplement: Feihe Investigational Formula
- Control Formula (Active Comparator): Control formula contains comparable macronutrients and micronutrients, but does not contain probiotics fortified with hydrolyzed whey protein
  Interventions: Dietary Supplement: Control Formula
- Breastfeeding (Other): breastmilk-feeding
  Interventions: Other: Breastfeeding

INTERVENTIONS:
Dietary Supplement: Feihe Investigational Formula — Participants in this arm will receive stage 1 and stage 2 Feihe investigational formulas. At the first (up to) 6 months, they will be fed with stage1 formula, and then switch to stage 2 formula until 12 months.
  Arms: Feihe Investigational Formula
Dietary Supplement: Control Formula — Participants in this arm will receive stage 1 and stage 2 Control formulas. At the first (up to) 6 months, they will be fed with stage1 formula, and then switch to stage 2 formula until 12 months.
  Arms: Control Formula
Other: Breastfeeding — Exclusively breastfed for the first 4 months and continue with supplement food without any marketed infant formula.
  Arms: Breastfeeding

SUMMARY:
The goal of this interventional clinical trial is to test the effectiveness of improving gut health in terms of frequency of bowel movements in newly born infants fed with Feihe investigational formula product containing probiotics fortified with hydrolyzed hey protein. The main question it aims to answer is:

- whether the frequency of bowel movements (through 12 months) of participants in the study product arm is significantly better than participants assigned in the other two arms.

240 qualified participants will be randomized to 3 arms (investigational formula, control formula, and breast-feeding) to consume assigned formula or breast-feeding for 12 months according to protocol. There will be up to 6 site visits arranged for each participant during the study, and all relevant clinical and questionnaire data, including the most important primary outcome - frequency of bowel movements through 12 months, will be captured, recorded and entered to CMTS (Clinical Management Trial System) for statistical analysis and reporting.

Researchers will compare the three arms to validate the assumption that the consumption of Feihe investigational formula product containing probiotics fortified with hydrolyzed hey protein will improve gut health in newly born infants, along with physical development.

ELIGIBILITY:
Inclusion Criteria:

* Newborn baby, study entry before weaning (within 28 days of birth)
* Exclusively formula fed for at least 3 days prior to study entry and plan to be exclusively formula fed during the study (formula groups) OR plan to be exclusively fed with human milk during the study (breastfeeding group).
* Gestational age of 37-42 weeks (36 weeks and six days is considered 36 weeks gestational age).
* Birth weight of 2500g (5 lbs. 8 oz.) to 4200g (9 lbs. 4 oz.).
* Signed informed consent obtained for infant's participation in the study.
* Parent or guardian of the infant agrees to not enroll the infant in another interventional clinical research study while participating in this study.

Exclusion Criteria:

* History of underlying metabolic or chronic disease; congenital malformation; or any other condition which, in the opinion of the Investigator, is likely to interfere with: the ability of the infant to ingest food, the normal growth and development of the infant, or the evaluation of the infant.
* Evidence of feeding difficulties or formula intolerance, such as vomiting or poor intake, at time of randomization (at investigator discretion).
* Evidence of growth problems or concern for growth.
* Infant was born large for gestational age (LGA) (defined as birth weight-for-age exceeding 90th percentile as plotted on the growth chart provided by Feihe) from mother who was diabetic at childbirth.
* Participant is immunocompromised (according to a doctor's diagnosis of immunodeficiency such as Combined Immunodeficiencies, DiGeorge Syndrome, Wiskott-Aldrich Syndrome, Severe Congenital Neutropenia and Secondary Immunodeficiencies linked to HIV infection, Down Syndrome or others) and children with known head/brain disease/injury.
* Use of probiotics/prebiotics before the study.

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 240 (Actual)
Dates: Start 2023-11-14 (Actual); Primary Completion 2025-04-03 (Actual); Study Completion 2025-04-03 (Actual)

PRIMARY OUTCOMES:
Stool Frequency | At the end of 12 months
  counting number of bowel movements per week, and adds together at the end of the study

SECONDARY OUTCOMES:
Stool Consistency | At the age of 15-28 days and 3, 6, 9, 12 months
  The rating score (0-5) of the stool consistency over the 24-hour period. The rating score of the stool consistency from the stool picture:
  0-No bowel movement;
  1. Hard- dry, hard pellets;
  2. Formed- definite shape, not dry;
  3. Soft-no definite shape, pasty;
  4. Unformed or seedy- no shape, some water or small lumps ;
  5. Waterly- no shape, mainly water where the score of 0-1 represents poor stool characteristics, while 2-5 represents fine stool characteristics.
Weight in grams | At the age of 15-28 days and 3, 6, 9, 12 months
  The weight measurement (gram) of the participant for each site visit
Height in cm | At the age of 15-28 days and 3, 6, 9, 12 months
  The height measurement (cm) of the participant for each site visit
Head circumference in cm | At the age of 15-28 days and 3, 6, 9, 12 months
  The head circumference measurement (cm) of the participant for each site visit
Amount of formula intake in ml | At the age of 15-28 days and 3, 6, 9, 12 months
  The 24-Hour dietary recall of Formula intake (amount in ml of study formula, any other infant formula or milk consumed) of the participant for each site visit
Medically-confirmed adverse events | baseline day to 12 months
  The frequency of medically-confirmed adverse events occurred during the study

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoyang Sheng, MD, Principal Investigator — School of Medicine, Shanghai Jiaotong University, Shanghai, China
Locations (3):
- China (3):
  - Jinhua Nanyuan Community Health Center, Jinhua, Zhejiang
  - Li Pu Community Hospital, Jinhua, Zhejiang
  - Qiu Bin Community Hospital, Jinhua, Zhejiang

IPD SHARING:
Plan to Share IPD: No